CLINICAL TRIAL: NCT02417558
Title: Study to Evaluate the Effectiveness of Personalized Brain Network Activation Technology in a Cognitive/Physical Computer-Game Blended Training of Elderly (Alterniity AR)
Brief Title: Cognitive/Physical Computer-Game Blended Training With Personalized Brain Network Activation Technology for the Elderly
Acronym: AlterniityAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: XtremeVRI AG (Industry)
Collaborators: Aristotle University Of Thessaloniki (Other); Greek Alzheimer's Association and Related Disorders (Other); Klinik Hirslanden, Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 84171-B
Record Dates: First submitted 2015-03-26; First posted 2015-04-15 (Estimated); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Mild Cognitive Impairment, So Stated; Mild Dementia; Healthy
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Alterniity Augmented Reality (AAR) (Experimental): AAR training Participants use the patent pending AAR exercise and gaming (exergaming) platform that combines a physical training component (PTC) and a cognitive training component (CTC) in closed-feedback loop with Personalized Brain Network Activity (PBNA) test from a portable EEG.
  Interventions: Behavioral: Alterniity Augmented Reality (AAR)
- Passive Control Participants (No Intervention): Passive Control Participants do not receive an intervention serving as passive controls
- Active (Active Comparator): Active Control Participants receive an alternative cognitive training scheme; software was built on purpose by the Aristotle University of Thessaloniki. The software is called VideoGrade and uses videos from Youtube (YouTube) documentaries (VideoGrade).
  Interventions: Behavioral: VideoGrade

INTERVENTIONS:
Behavioral: Alterniity Augmented Reality (AAR) — AAR is a patent pending exercise and gaming (exergaming) computer platform with a physical training component (PTC) and a cognitive training component (CTC). It fully immerses a user inside a virtual environment where he is practising complex everyday activities, such as going shopping, using the transportation, visiting a foreign city, eating at a restaurant, cooking dinner etc. His motor behaviour is monitored by means of motion capture, while immersed at this full-body immersion. In addition his cognition is monitored in real-time with Personalized Brain Network Activity (PBNA) screening. Both the motor and brain analyses are then used to update the configuration, type and difficulty of the AAR scenarios.
  Other Names: VR-DOT; VPH-DARE@IT
  Arms: Alterniity Augmented Reality (AAR)
Behavioral: VideoGrade — Active cognitive training by use of the VideoGrade software by Aristotle University of Thessaloniki.
  Arms: Active

SUMMARY:
The study involves a novel Virtual Reality Interface that offers full-body immersion "Alterniity AR" and more specifically computer exercises blended with game activities. It was hypothesized that "Alterniity AR" facilitated, game blended cognitive and/or physical exercise improves global cognition when compared to control groups; moreover, these improvements may be manifested by brain activity changes. The investigators explore here the impact of potential moderators on combined exercise-induced cognitive benefits, as well as, individual/separate training schemes.

In addition, the proposed study will provide Alterniity AR" in a closed feedback loop with a direct, reliable, and non-invasive method for assessing changes in brain activity associated with elderly in risk of dementia. The paradigm for the current study will combine neurophysiological knowledge with mathematical signal processing and pattern recognition methods to temporally and spatially map brain function, connectivity and synchronization.

DETAILED DESCRIPTION:
Currently, there is no direct, reliable, bed-side, and non-invasive method for assessing changes in brain activity associated with elderly in risk of dementia. Event Related Potentials (ERPs), which are temporal reflections of the neural mass electrical activity of cells in specific regions of the brain that occur in response to stimuli, may offer such a method, as they provide both a noninvasive and portable measure of brain function. The ERPs provide excellent temporal information, but spatial resolution for ERPs has traditionally been limited. However, by using high-density electroencephalograph (EEG) recording spatial resolution for ERPs is improved significantly. The proposed study will provide additional evidence for the utility and contribution of a Personalized Brain Network Activation (PBNA) test (reflecting temporal and spatial changes in brain activity as well as brain functional connectivity associated with minor neurocognitive disorder) in early dementia management.

The study is conducted in 2 sites: Switzerland and Greece. It uses a pre-post-test design with the between-participant factor group [intervention(s) vs. passive and/or active control]. Post-test will be conducted within 2 weeks after completion of the exercise period. Interventions will be carried out within day care centres, hospitals, senior care centres, a memory outpatient centre, local parishes, and at participants' homes. Centres will provide 8-12 exercise weeks per year for 3 years, with a frequency of at least 3 "Alterniity AR" sessions per week, resulting in at least 24-36 intervention sessions each year of the study. The closed feedback loop with a direct PBNA test is basically divided to 3 phases - first EEG data is collected from subjects using a portable EEG system while the participants are performing the "Alterniity AR" intervention. The EEG data is then analysed offline. Finally, the "Alterniity AR" exercise type, configuration and difficulty level is updated based on the analysed data.

The Greek site population (n=581) in majority subjects with mild cognitive impairment (MCI) has been described before with Clinical Trial Registration: NCT02313935

The Swiss population (n=126) was 20 healthy controls (HC), 20 mild to moderate Alzheimer's disease (AD) patients, 20 vascular dementia (VAD) patients, 20 fronto-temporal dementia (FTD) patients and 40 subjects with mild cognitive impairment (MCI). This population has been previously described at the following ClinicalTrials.gov Identifier: NCT02050464.

ELIGIBILITY:
Inclusion Criteria:

* no severe cognitive impairment measured by Mini-Mental State Examination (MMSE) ≥ 18
* fluent language skills
* agreement of a medical doctor
* time commitment to the test and exercise protocol.

Exclusion Criteria:

* concurrent participation in another study
* severe physical or psychological disorders which precluded participation in the intervention (i.e., inability to follow instructions)
* unrecovered neurological disorders such as stroke, traumatic brain injury, unstable medication within the past three months
* severe and uncorrectable vision problems, or hearing aid for less than three months.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 607 (Actual)
Dates: Start 2015-02; Primary Completion 2018-09 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Change in Diagnostic Area Under the Receiver Operating Characteristic Curve (ROC-AUC) | baseline to 40 months
  The Digital Neuro Signatures (DNS) score will be tested in this prospective cohort. Sensitivity, specificity and accuracy of the DNS score will be tested for detecting intervention responses for both the placebo and the study groups and will be compared to the intervention responses measured by the neuropsychological test battery.

SECONDARY OUTCOMES:
Physical Fitness | 2 months / 6+2 months / 12+2 months
  Physical capacity was measured by means of the Senior Fitness Test
Episodic memory | 2 months / 6+2 months / 12+2 months
  calculated by averaging z-standardized sub-scores of the three cognitive tests (CVLT, the Digit Span Test and TMT).
Working Memory | 2 months / 6+2 months / 12+2 months
  calculated by averaging z-standardized sub-scores of the three cognitive tests (CVLT, the Digit Span Test and TMT).
Executive Function | 2 months / 6+2 months / 12+2 months
  calculated by averaging z-standardized sub-scores of the three cognitive tests (CVLT, the Digit Span Test and TMT).
World Health Organization Quality of Life (WHOQoL) | 2 months / 6+2 months / 12+2 months
  The World Health Organization Quality of Life (WHOQOL-100) questionnaire is a generic quality of life (QoL) measurement tool used in various cultural and social settings and across different patient and healthy populations. It was developed collaboratively in 15 cultural settings over several years and has been field tested in 37 centres. It consists of 100-questions that has been translated into 29 languages. It yields a multi-dimensional profile of scores across domains and sub-domains (facets) of quality of life. More recently, the WHOQOL-BREF, an abbreviated 26 item version has been developed. Domains/dimensions 6: Physical, psychological, level of independence, social relationships, environment, spirituality/religion/personal beliefs
Instrumental Activities of daily living | 2 months / 6+2 months / 12+2 months
  instrumental activities of daily living (IADL)
Depressive symptoms | 2 months / 6+2 months / 12+2 months
  Geriatric Depression Scale (GDS)
Overall brain function | 12 months
  The paradigm for the current study will combine neurophysiological knowledge with mathematical signal processing and pattern recognition methods to temporally and spatially map brain function, connectivity and synchronization.
Verbal learning and memory as assessed using California Verbal Learning Test (CVLT) | 2 months / 6+2 months / 12+2 months
  California Verbal Learning Test (CVLT) used to assess verbal learning and memory
Verbal short-term memory as assessed using the Digit Span Test | 2 months / 6+2 months / 12+2 months
  Digit Span Test and the Trail Making Test (TMT) used to assess verbal short-term memory

CONTACTS AND LOCATIONS:
Overall Officials: Magda Tsolaki, PhD, Study Director — GAADRD

REFERENCES:
- [Background] Tarnanas I. A virtual environment for the assessment and the rehabilitation of the visuo-constructional ability in dementia patients. Stud Health Technol Inform. 2000;70:341-3. PMID 10977568
- [Background] Tarnanas I, Schlee W, Tsolaki M, Muri R, Mosimann U, Nef T. Ecological validity of virtual reality daily living activities screening for early dementia: longitudinal study. JMIR Serious Games. 2013 Aug 6;1(1):e1. doi: 10.2196/games.2778. PMID 25658491
- [Background] Laskaris NA, Tarnanas I, Tsolaki MN, Vlaikidis N, Karlovasitou AK. Improved detection of amnestic MCI by means of discriminative vector quantization of single-trial cognitive ERP responses. J Neurosci Methods. 2013 Jan 30;212(2):344-54. doi: 10.1016/j.jneumeth.2012.10.014. Epub 2012 Nov 9. PMID 23147007
- [Background] Tarnanas I, Tsolaki M, Nef T, M Muri R, Mosimann UP. Can a novel computerized cognitive screening test provide additional information for early detection of Alzheimer's disease? Alzheimers Dement. 2014 Nov;10(6):790-8. doi: 10.1016/j.jalz.2014.01.002. Epub 2014 Mar 18. PMID 24656838
- [Background] Tarnanas I, Laskaris N, Tsolaki M, Muri R, Nef T, Mosimann UP. On the comparison of a novel serious game and electroencephalography biomarkers for early dementia screening. Adv Exp Med Biol. 2015;821:63-77. doi: 10.1007/978-3-319-08939-3_11. PMID 25416111
- See also: Assessing Virtual Reality Environments as Cognitive Stimulation Method for Patients with Mild Cognitive Impairment (MCI) — http://link.springer.com/chapter/10.1007/978-3-642-45432-5_4